CLINICAL TRIAL: NCT06109051
Title: EndeavorOTC™ Prospective Product Registry
Status: Active, not recruiting | Type: Observational
Sponsor: Akili Interactive Labs, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Akili-065
Record Dates: First submitted 2023-10-23; First posted 2023-10-31 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- EndeavorOTC Users: All users who subscribe to EndeavorOTC for any duration
  Interventions: Device: EndeavorOTC

INTERVENTIONS:
Device: EndeavorOTC — EndeavorOTC™ is an over-the-counter digital therapeutic designed to improve attention function, ADHD symptoms, and quality of life in users 18 years of age and older with primarily inattentive or combined-type ADHD, who have been identified as having a significant attentional impairment. EndeavorOTC utilizes the same proprietary technology underlying EndeavorRx, a prescription digital therapeutic indicated to improve attention function in children ages 8-12. EndeavorOTC is not intended to be a replacement for any form of ongoing treatment. EndeavorOTC is deployed on mobile devices and incorporates adaptive, simultaneous cognitive tasks in a consumer-grade action videogame-based platform with high-quality graphics and reward mechanisms.
  Other Names: AKL-T01A

SUMMARY:
The EndeavorOTC product registry aims to collect real world data from EndeavorOTC users. The objectives of this registry are to describe clinical and demographic characteristics, treatment patterns, clinical and quality of life outcomes, and healthcare utilization in EndeavorOTC users in a real-world setting.

DETAILED DESCRIPTION:
All EndeavorOTC users who subscribe to EndeavorOTC are invited to participate in this product registry. Users must provide their informed consent and have an active subscription to the product at time of enrollment to participate. Study activities are emailed to participants at baseline, 1, 2, 3, 6, 9, and 12-months after enrollment. Study activities consist of an online survey and online ADHD assessment. All data are captured electronically and securely through commercial data capture platforms.

ELIGIBILITY:
Inclusion Criteria:

* Has an active EndeavorOTC™subscription
* Provide informed consent to participate in the registry

Exclusion Criteria:

* N/A

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: EndeavorOTC users may enroll and participate in the product registry for the full year regardless of the length of their EndeavorOTC subscription.
Sampling Method: Non-Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Computerized Adaptive Test, Mental Health (CAT-MH®) | Baseline, Months 1, 2, 3, 6, 9, 12
  Computerized Adaptive Test, Mental Health (CAT-MH®) is a distinct suite of computer adaptive tests that is based on multidimensional item response theory. The adult ADHD module is a dimensional severity measure of attention-deficit/hyperactivity disorder symptomatology for adults 18 and over. The number and selection of questions within the assessment varies as individuals' initial item responses are used to determine a provisional estimate of their standing on the measured trait to be used for subsequent item selection. Items are scored on a Likert scale of 1 (Not at all), 2 (Just a little), 3 (Somewhat), 4 (Quite a bit), and 5 (Very much).
  Negative change in score indicates improvement in ADHD severity.
Conners' Adult ADHD Rating Scales-Self Report: Short Version (CAARS-S:S) | Baseline, Months 1, 2, 3, 6, 9, 12
  Conners' Adult ADHD Rating Scales-Self Report: Short Version (CAARS-S:S) provides an assessment of symptoms and behaviors associated with ADHD in adults ages 18 and older. The short versions of the self-report form (CAARS-S:S) contain 26 items that are scored on a scale of 0 (Not at all, never), 1 (Just a little, once in a while), 2 (Pretty much, often), and 3 (Very much, very frequently).
  Negative change in score indicates improvement in ADHD symptoms and behaviors.
Adult ADHD Quality of Life (AAQoL) | Baseline, Months 1, 2, 3, 6, 9, 12
  Adult ADHD Quality of Life (AAQoL) is a 29-item, self-report measure of functioning in a variety of life domains and adult roles. Items are rated on a 5-point scale that are transformed into a 0-100 scale, with higher scores reflecting higher quality of life. Scores are calculated for life productivity, psychological health, life outlook, and relationships, in addition to total score.
  Positive change in score indicates improvement in quality of life.
Patient Health Questionnaire - 4 items (PHQ-4) | Baseline, Months 1, 2, 3, 6, 9, 12
  Patient Health Questionnaire - 4 items (PHQ-4) is an ultra-brief, validated screening assessment for anxiety and depression, consisting of four-items that are scored on a Likert scale of 0 (not at all), 1 (several days), 2 (more than half the days), and 3 (nearly every day). A higher score indicates greater levels of depression and anxiety.
  Negative change in score indicates improvement in anxiety and depression.
Treatment Inventory of Costs in Patients with psychiatric disorders (TIC-P) | Baseline, Months 3, 6, 9, 12
  Treatment Inventory of Costs in Patients with psychiatric disorders (TIC-P) is a questionnaire that assesses the utilization of medical care and productivity loss. Select questions from the TIC-P questionnaire will be used to estimate costs of healthcare utilization. This assessment will be administered once every 3 months. Participants are asked to provide the number of appointments they have had with a specific healthcare provider or service in the past three months. The sum of total number of appointments utilized within a three month period will be compared between study time points.
  Negative change in total number of appointments indicates improvement.
Percent work time missed due to ADHD, as measured by Work Productivity and Activity Impairment Questionnaire plus Classroom Impairment Questions: Specific Health Problem (WPAI+CIQ:SHP), Version 2.0 | Baseline, Months 1, 2, 3, 6, 9, 12
  Work Productivity and Activity Impairment Questionnaire plus Classroom Impairment Questions: Specific Health Problem (WPAI+CIQ:SHP), Version 2.0 is a 10-item, validated self-report questionnaire which is based on an individual's absenteeism, presenteeism, work or classroom productivity loss, and activity impairment due to a specific disease/condition. This questionnaire has been adapted to the specific health problem of ADHD. Outcomes are expressed as impairment percentages (0-100), with higher numbers indicating greater impairment and less productivity.
  Negative change indicates improvement.
Percent impairment while working due to ADHD, as measured by WPAI+CIQ:ADHD | Baseline, Months 1, 2, 3, 6, 9, 12
  Work Productivity and Activity Impairment Questionnaire plus Classroom Impairment Questions: Specific Health Problem (WPAI+CIQ:SHP), Version 2.0 is a 10-item, validated self-report questionnaire which is based on an individual's absenteeism, presenteeism, work or classroom productivity loss, and activity impairment due to a specific disease/condition. This questionnaire has been adapted to the specific health problem of ADHD. Outcomes are expressed as impairment percentages (0-100), with higher numbers indicating greater impairment and less productivity.
  Negative change indicates improvement.
Percent overall work impairment due to ADHD, as measured by WPAI+CIQ:ADHD | Baseline, Months 1, 2, 3, 6, 9, 12
  Work Productivity and Activity Impairment Questionnaire plus Classroom Impairment Questions: Specific Health Problem (WPAI+CIQ:SHP), Version 2.0 is a 10-item, validated self-report questionnaire which is based on an individual's absenteeism, presenteeism, work or classroom productivity loss, and activity impairment due to a specific disease/condition. This questionnaire has been adapted to the specific health problem of ADHD. Outcomes are expressed as impairment percentages (0-100), with higher numbers indicating greater impairment and less productivity.
  Negative change indicates improvement.
Percent class time missed due to ADHD, as measured by WPAI+CIQ:ADHD | Baseline, Months 1, 2, 3, 6, 9, 12
  Work Productivity and Activity Impairment Questionnaire plus Classroom Impairment Questions: Specific Health Problem (WPAI+CIQ:SHP), Version 2.0 is a 10-item, validated self-report questionnaire which is based on an individual's absenteeism, presenteeism, work or classroom productivity loss, and activity impairment due to a specific disease/condition. This questionnaire has been adapted to the specific health problem of ADHD. Outcomes are expressed as impairment percentages (0-100), with higher numbers indicating greater impairment and less productivity.
  Negative change indicates improvement.
Percent overall classroom impairment due to ADHD, as measured by WPAI+CIQ:ADHD | Baseline, Months 1, 2, 3, 6, 9, 12
  Work Productivity and Activity Impairment Questionnaire plus Classroom Impairment Questions: Specific Health Problem (WPAI+CIQ:SHP), Version 2.0 is a 10-item, validated self-report questionnaire which is based on an individual's absenteeism, presenteeism, work or classroom productivity loss, and activity impairment due to a specific disease/condition. This questionnaire has been adapted to the specific health problem of ADHD. Outcomes are expressed as impairment percentages (0-100), with higher numbers indicating greater impairment and less productivity.
  Negative change indicates improvement.
Percent activity impairment due to ADHD, as measured by WPAI+CIQ:ADHD | Baseline, Months 1, 2, 3, 6, 9, 12
  Work Productivity and Activity Impairment Questionnaire plus Classroom Impairment Questions: Specific Health Problem (WPAI+CIQ:SHP), Version 2.0 is a 10-item, validated self-report questionnaire which is based on an individual's absenteeism, presenteeism, work or classroom productivity loss, and activity impairment due to a specific disease/condition. This questionnaire has been adapted to the specific health problem of ADHD. Outcomes are expressed as impairment percentages (0-100), with higher numbers indicating greater impairment and less productivity.
  Negative change indicates improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Scott H Kollins, PhD, Principal Investigator — Akili Interactive Labs, Inc.
Locations (1):
- Akili Interactive Labs, Inc., Boston, Massachusetts, United States